CLINICAL TRIAL: NCT01860534
Title: "Eye Protection After Mydriatic Use for ROP Screening: Impact on Vitals Signs and Pain Scores"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-039
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2014-05

CONDITIONS: Light Sensitivity
Keywords: pain; mydriasis; light
MeSH Terms: conditions — Photophobia; Pain; Mydriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eye patches covers (Experimental): The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam while group B was unpatched for their first ROP exam and patched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
  Interventions: Behavioral: eye covers
- no eye patches covers (No Intervention): The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam while group B was unpatched for their first ROP exam and patched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.

INTERVENTIONS:
Behavioral: eye covers — The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam while group B was unpatched for their first ROP exam and unpatched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
  Other Names: eye patches (Natus biliband)
  Arms: Eye patches covers

SUMMARY:
Pupillary dilation induced by mydriatic agents during Retinopathy of Prematurity exams can persist for hours. Despite regular use of eye protection for mydriatic-induced light sensitivity for infants, children and adults, eye protection after mydriasis has not been addressed in neonates. This study examines the use of eye patches to protect the dilated pupil from light exposure and their impact on vital signs and pain scores. prevents tachycardia, tachypnea and discomfort in neonates after ROP screening.

DETAILED DESCRIPTION:
Pain management for Retinopathy of prematurity (ROP) screening focuses on pharmacological and non-pharmacological interventions during the actual eye examination. Management of pain related to increased light sensitivity during the post-mydriasis period has not been described.

This prospective, randomized study evaluated the impact of protecting the eyes from ambient light exposure post mydriasis. Vital signs and pain scales were recorded in infants randomized to either wear or not wear eye patches after mydriasis for their ROP exam. Infants less than 30 weeks gestational age or less than 1500 grams at birth were included. Standard statistical methods were used to compare vital signs and pain scores for each group at baseline, 1 and 3 hours after mydriasis.

ELIGIBILITY:
Inclusion Criteria:

* All infants with gestational age at birth of 30 weeks or less or with birth weight less than 1500g undergoing their first ROP exam in the Infant Special Care Unit (ISCU) at UTMB.

Exclusion Criteria:

* Infants were excluded if they had any congenital malformation or syndrome; a history of eye surgery or were receiving inotropics medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika M. Espino-Torres, MD, Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2011 to september 2012. At the University of Texas medical Branch.
Pre-assignment Details: 60 neonates were excluded prior to randomization since they did not meet inclusion criteria, refused to participate or other reasons.
Groups:
- Eye Patch Initially Then no Eye Patch: The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care. Two groups were created to ensure comparison of similar gestational ages at the time of initial and secondary exams as younger neonates are often more ill. This added control was to minimize confounding by age or illness.
- no Eye Patches Initially Then Eye Patches: The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group B was unpatched for their first ROP exam and patched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care. Two groups were created to ensure comparison of similar gestational ages at the time of initial and secondary exams as younger neonates are often more ill. This added control was to minimize confounding by age or illness.
Period: ROP #1
Arm/Group | Eye Patch Initially Then no Eye Patch | no Eye Patches Initially Then Eye Patches
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Needed treatment for ROP | 0 | 1
Period: ROP #2
Arm/Group | Eye Patch Initially Then no Eye Patch | no Eye Patches Initially Then Eye Patches
Started | 14 | 13
Completed | 13 | 13
Not Completed | 1 | 0
Not completed — discharged prior to ROP #2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Eye Patches Initially Then no Patches: The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
- no Eye Patches Initially Then Eye Patches: The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group B was unpatched for their first ROP exam and patched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
- Total: Total of all reporting groups
Arm/Group | Eye Patches Initially Then no Patches | no Eye Patches Initially Then Eye Patches | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.54 (0.04) | 0.53 (0.04) | 0.53 (0.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: At 3 times (pre-mydriasis, 1 hour and 3 hours after Cyclomydril drops), subjects were exposed to ambient lighting for a period of five minutes. This usually entailed removing isolette covers and exposing the patient to the ambient room light. During this time, pain and vital signs were recorded every minute. Heart rate was recorded directly from their cardio-respiratory monitor (Agilent M1106C). The mean of the five recorded values for each variable was used
Time Frame: pre-mydriasis, 1 hour and 3 hours after mydriatic drops
Measure: Mean (Standard Deviation); unit: Beats per minutes
Groups:
- Eye Patches Covers (ROP #1 and ROP #2); no Eye Patches Covers (ROP #1 and ROP #2): The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam while group B was unpatched for their first ROP exam and unpatched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
Arm/Group | Eye Patches Covers (ROP #1 and ROP #2) | no Eye Patches Covers (ROP #1 and ROP #2)
Number analyzed (Participants) | 26 | 26
Beats per minutes
  Baseline | 154 (8) | 154 (12)
  1 hour post dilation | 152 (8) | 163 (10)
  3 hour post dilation | 154 (8) | 164 (9)

2. Secondary Outcome: Respiratory Rate
Description: At 3 times (pre-mydriasis, 1 hour and 3 hours after Cyclomydril drops), subjects were exposed to ambient lighting for a period of five minutes. This usually entailed removing isolette covers and exposing the patient to the ambient room light. During this time, pain and vital signs were recorded every minute. Respiratory rate was recorded directly from their cardio-respiratory monitor (Agilent M1106C). The mean of the five recorded values for each variable was used
Time Frame: pre-mydriasis, 1 hour and 3 hours after mydriatic drops
Measure: Mean (Standard Deviation); unit: Breaths per minutes
Groups:
- Eye Patches Covers; no Eye Patches Covers: The infants were randomly assigned by alternating enrolled patients between one of two groups prior to their first ROP screening. Group A was patched for their first ROP exam and then unpatched for their second exam while group B was unpatched for their first ROP exam and unpatched for their second exam. The patched subjects had eye covers after their eyes were dilated, and the unpatched subjects had comfort measures similar to the patched subjects but their eyes were not covered. The patching of the eyes was done in the same way that it is done for eye protection during phototherapy, with the same model of eye patches (Natus biliband) and with the same nursing care.
Arm/Group | Eye Patches Covers | no Eye Patches Covers
Number analyzed (Participants) | 26 | 26
Breaths per minutes
  Baseline | 54 (13) | 47 (8)
  1 hour post dilation | 54 (13) | 52 (13)
  3 hour post dilation | 55 (11) | 50 (10)

3. Secondary Outcome: Oxygen Percent Saturation
Description: At 3 times (pre-mydriasis, 1 hour and 3 hours after Cyclomydril drops), subjects were exposed to ambient lighting for a period of five minutes. This usually entailed removing isolette covers and exposing the patient to the ambient room light. During this time, pain and vital signs were recorded every minute. Oxygen percent saturation was recorded directly from their cardio-respiratory monitor (Agilent M1106C). The mean of the five recorded values for each variable was used
Time Frame: pre-mydriasis, 1 hour and 3 hours after mydriatic drops
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Eye Patches Covers | no Eye Patches Covers
Number analyzed (Participants) | 26 | 26
percent saturation
  Baseline | 98 (3) | 98 (3)
  1 hour post dilation | 98 (3) | 98 (3)
  3 hour post dilation | 98 (3) | 98 (2)

4. Secondary Outcome: Pain
Description: At 3 times (pre-mydriasis, 1 hour and 3 hours after Cyclomydril drops), subjects were exposed to ambient lighting for a period of five minutes. This usually entailed removing isolette covers and exposing the patient to the ambient room light. During this time, pain and vital signs were recorded every minute. Pain scores were recorded by direct observation using the Neonatal and Infant Pain Scale (NIPS). The mean of the five recorded values for each variable was used. NIPS scoring consists of 6 measures associated with neonatal or infant pain, each with a range of 0-7 with low scores (0-2) associated with no pain and scores > to 4 associated with severe pain. Maximum scoring would be 42 for severe pain and minimal being 0 for no pain. The six measures on NIPS include: facial expression, crying, breathing patterns, arm movements, leg movements and state of arousal.
Time Frame: pre-mydriasis, 1 hour and 3 hours after mydriatic drops
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eye Patches Covers | no Eye Patches Covers
Number analyzed (Participants) | 26 | 26
units on a scale
  Baseline | 0.4 (0.3) | 0.3 (0.5)
  1 hour post dilation | 0.1 (0.2) | 1.1 (0.7)
  3 hour post dilation | 0.2 (0.2) | 1 (0.6)

ADVERSE EVENTS:
Arm/Group | Eye Patches Covers | no Eye Patches Covers
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No